CLINICAL TRIAL: NCT04769388
Title: The Efficacy and Safety of Osimertinib Plus Carboplatin and Pemetrexed Versus Osimertinib Monotherapy in Metastatic EGFRm NSCLC Patients With EGFRm Persistence in ctDNA at 3 Weeks After 1L Osimertinib: A Multicenter, Randomized Controlled Study
Brief Title: Osimertinib Plus Chemotherapy vs Osimertinib in EGFRm NSCLC With Persistence Week-3 ctDNA EGFRm After 1L Osimertinib
Acronym: FLAME
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Cancer Prevention & Treatment Society (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-19-20439
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osimertinib 80 mg QD and platinum-based chemotherapy (Experimental): Osimertinib 80 mg in combination with pemetrexed (500 mg/m2) plus carboplatin (AUC5) on Day 1 of 21day cycles (every 3 weeks) for up to 6 cycles, followed by Osimertinib daily with pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Interventions: Drug: Osimertinib; Drug: Pemetrexed/Carboplatin
- Osimertinib 80mg QD (Active Comparator): All patients randomized into this will only receive Osimertinib 80mg.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Pemetrexed (500 mg/m2) plus carboplatin (AUC5) on Day 1 of 21day cycles (every 3 weeks) for up to 6 cycles, followed by Osimertinib daily with pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Other Names: AZD9291; Tagrisso
Drug: Pemetrexed/Carboplatin — Pemetrexed (500 mg/m2) plus carboplatin (AUC5) on Day 1 of 21day cycles (every 3 weeks) for up to 6 cycles, followed by Osimertinib daily with pemetrexed maintenance (500 mg/m2) every 3 weeks.
  Arms: Osimertinib 80 mg QD and platinum-based chemotherapy

SUMMARY:
This is a prospective, randomised, open-label, positive-controlled study to investigate the efficacy and safety of Osimertinib plus Carboplatin/Pemetrexed versus Osimertinib monotherapy in metastatic EGFRm NSCLC patients with EGFRm persistence in ctDNA at 3 weeks after first-line therapy with Osimertinib.

ELIGIBILITY:
Inclusion Criteria:

* Provision and signed of informed consent prior to any study specific procedures;
* Male or female, aged at least 18 years;
* Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1;
* Newly diagnosed, and histologically documented metastatic non-squamous NSCLC with sensitizing EGFR mutations positive, and classified as stage IV or recurrent NSCLC which are not amenable to curative surgery or radiotherapy;
* Life expectancy of at least 3 months at recruitment;
* Only the patients receiving osimertinib as 1L treatment and meeting the following criteria will be considered:

A. Prior to 1L osimertinib:

1. History of EGFRm (exon 19 deletion or exon 21 L858R) in the plasma ctDNA by the local testing methods.
2. No previous systemic treatment. Adjuvant therapies, or definitive radiation/chemoradiation are permitted as long as treatment was completed at least 6 months prior to receiving 1L treatment.
3. Patients with asymptomatic and stable CNS metastases for at least 2 weeks will be allowed, including leptomeningeal metastases.

B. Prior to randomization: Patients after 3 weeks of 1L osimertinib treatment who have persistence ctDNA EGFRm by SuperARMS at 3 weeks will be considered to be enrolled. They will need to further meet the criteria below before randomization:

1. Patients without disease progression by RECIST 1.1 evaluation;
2. At least 1 measurable extracranial lesion according to RECIST 1.1 .
3. Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential.
4. Male subjects should be willing to agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study;
* History of hypersensitivity to active or inactive excipients of Osimertinib and/or Pemetrexed and/or Carboplatin or drugs with a similar chemical structure or class to Osimertinib and/or Pemetrexed and/or Carboplatin;
* For patients, inability to collect plasma samples at baseline and disease progression;
* QT prolongation or any clinically important abnormalities in rhythm;
* Any evidence of severe or uncontrolled systemic diseases;
* Currently receiving medications or herbal supplements known to be strong inducers of CYP3A4;
* Any unresolved toxicities from prior therapy greater than CTCAE 5.0 grade 1 at the time of starting study treatment.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
* Inadequate bone marrow reserve or organ function;
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Contraindication for osimertinib, pemetrexed and carboplatin according to China approved label.
* Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | The primary analysis of Progression-free survival (PFS) based on investigator assessment will occur when PFS maturity is observed at approximately 30 months after the first patient is randomized.
  Progression-free survival (PFS) using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
OS rate at 18 months | The OS rate at 18 months will be defined as the Kaplan-Meier estimate of OS at 18 months.
  Proportion of patients alive at 18 months
Objective Response Rate (ORR) | Objective Response Rate analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 30 months from the first patient being randomized.
  ORR (per RECIST 1.1 using Investigator assessments) is defined as the number (percent) of patients with at least 1 visit response of CR or PR.
Disease Control Rate (DCR) | Disease control rate analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 30 months from the first patient being randomized.
  Disease control rate (DCR) is defined as the percentage of subjects who have a best overall response of CR or PR or SD by RECIST 1.1 as assessed by the Investigator.
Duration of Response (DoR) | Duration of Response analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 30 months from the first patient being randomized.
  DoR is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Depth of Response | Depth of Response analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 30 months from the first patient being randomized.
  Depth of response by Investigator is defined as the relative change in the sum of the longest diameters of RECIST target lesions at the nadir in the absence of NLs or progression of NTLs when compared to baseline.
Safety and tolerability: Adverse event | Safety and tolerability analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 30 months from the first patient being randomized.
  All Adverse events/≥grade 3 AE/SAE incidence rate (AE/SAE graded by CTCAE v5); All ADR incidence rate; AESI: ILD/pneumonitis-like event, Cardiac failure
Molecular resistance mechanism | Molecular resistance mechanism analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 30 months from the first patient being randomized.
  To evaluate potential molecular resistance mechanism by biomarker analysis of plasma at baseline and disease progression and tissue samples (if applicable) by next-generation sequencing (NGS).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No